CLINICAL TRIAL: NCT01617863
Title: Central Hemodynamics, Arterial Stiffness, Heartrate and Endothelial Dysfunktion During the European Soccer Championship 2012
Brief Title: Hemodynamics During the Soccer Championship 2012
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Collaborators: Universitätsklinikum Greifswald, Greifswald, Mecklenburg-Vorpommern, Germany (Unknown); Universitätsklinikum Erlangen, Erlangen, Bayern, Germany (Unknown); Universitätsklinikum Eppendedorf, Hamburg, Germany (Unknown); UKSH Campus Kiel, Kiel, Germany (Unknown)
Responsible Party: Principal Investigator, PD. Dr. med Michael Reppel, PD Dr. med Reppel, University Hospital Schleswig-Holstein
Other Study IDs: HL-Med2-EM-2012
Record Dates: First submitted 2012-06-08; First posted 2012-06-12 (Estimated); Last update posted 2012-07-03 (Estimated); Status verified 2012-06

CONDITIONS: Severe Cardiomyopathy; Angina, Unstable; Myocardial Infarction; Angina, Stable
MeSH Terms: conditions — Cardiomyopathies; Angina, Unstable; Myocardial Infarction; Angina, Stable

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — EDTA-Blood, Serum
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to determine in soccer fans whether and to which extend positive or negative emotions during the European soccer Championship affects Central Hemodynamics, Arterial Stiffness, Heartrate and Endothelial Dysfunktion.

ELIGIBILITY:
Inclusion Criteria:

Best fit:

* cardiomyopathy "severe myocardial disease leading to heart failure"
* Angina, stable for at least 7 days
* Myocardial infarction during 4 weeks before inclusion, actually stable condition
* Angina, Stable, CCS II-IV

Exclusion Criteria:

* not interested in soccer championship
* age <18y
* dementia
* atrial tachycardia
* drug/alcohol abuse
* chronic kidney disease, stage 5
* pulmonary/tricuspid valve insufficiency/stenoses
* non compliant

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic, clinical employees, students
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2012-06; Primary Completion 2012-07 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Reppel, PD. Dr. med, Study Director — UKSH- Lübeck Medizinische Klinik 2
Locations (4):
- Germany (4):
  - Universitätsklinikum Erlangen, Erlangen, Bavaria
  - Universitätsklinikum Eppendorf, Hamburg, Hamburg
  - Universitätsklinikum Greifswald, Greifswald, Mecklenburg-Vorpommern
  - UKSH-Lübeck, Lübeck, Schleswig-Holstein